CLINICAL TRIAL: NCT00351494
Title: Myoma Microvascularization Analysis Using Sonovue Before and After Uterine Artery Embolization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Other Study IDs: HP06-HM/FIBROME
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Myoma
Keywords: embolization; contrast enhanced ultrasound; myoma; uterine artery; microvascularisation
MeSH Terms: conditions — Myoma | interventions — Embolization, Therapeutic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: contrast enhanced ultrasonography — Three contrast-enhanced ultrasonography : before embolization, after one day and after 6 months.
  Abdominal route 2.4 ml sonovue per injection / bolus
Procedure: embolization — Intervention is described in the case report form for each patient

SUMMARY:
Contrast-enhanced ultrasound is supposed to improve the detection of myomas as well as improve the follow-up after specific treatments like embolization. It will also help the investigators better understand the mechanism of success or failure for embolization and could reduce the amount of particles injected by determining the endpoint of the procedure in order to treat the myomas while preserving the myometrium.

DETAILED DESCRIPTION:
Before embolization of the uterine artery, 40 patients with unique or multiple myomas will be included prospectively in our study and evaluated with sonography before and after injection of Sonovue (2.4 ml) (Bracco Int Milano Italy). Pelvic ultrasound with contrast enhancement will be done the day after and six months after the procedure.

Microvascularization of the myomas and the endometrium will be described. Some tiny myomas which are not visible on conventional sonography could be identified for a perfect matching with MRI detection.

ELIGIBILITY:
Inclusion Criteria:

* Uterine myomas with solid tissue (greater diameter lower than 15 cm)
* The embolization is planified during the 15 days after the contrast ultrasonography
* Written informed consent is signed

Exclusion Criteria:

* Intracavitary uterine mass possibly due to a polyp or endometrial cancer
* Necessity of using the endovaginal way of ultrasonography because of the myoma's size and accessibility
* Menopause
* Pregnancy and breastfeeding
* Recent cardiac affection
* History of acute cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women candidate for embolization of myomas
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To investigate the usefulness of contrast-enhanced ultrasound with real-time imaging technique in the assessment of vascular patterns from myomas myometrium and ovaries before and after uterine artery embolization | Inclusion period and follow-up

SECONDARY OUTCOMES:
Accordance between contrast-enhanced imaging and IRM | inclusion period and follow-up
Accordance between early vascular patterns due to embolization of the fibroma and the success of the technique which is evaluated after 6 month | inclusion period and follow-up
Relationship between the post embolization pain and the vascular change of the fibroma and the myometrium | inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Henri MARRET, Pr, Principal Investigator — Service de Gynécologie Obstétrique CHRU TOURS; François TRANQUART, Pr, Study Director — Centre d'Innovation Technologique CHRU TOURS
Locations (1):
- Centre d'Innovation Technologique-Ultrasons, Tours, France

REFERENCES:
- [Background] Tranquart F, Brunereau L, Cottier JP, Marret H, Gallas S, Lebrun JL, Body G, Herbreteau D, Pourcelot L. Prospective sonographic assessment of uterine artery embolization for the treatment of fibroids. Ultrasound Obstet Gynecol. 2002 Jan;19(1):81-7. doi: 10.1046/j.0960-7692.2001.00535.x. PMID 11851974
- [Background] Marret H, Cottier JP, Alonso AM, Giraudeau B, Body G, Herbreteau D. Predictive factors for fibroids recurrence after uterine artery embolisation. BJOG. 2005 Apr;112(4):461-5. doi: 10.1111/j.1471-0528.2004.00487.x. PMID 15777445
- [Background] Marret H, Tranquart F, Sauget S, Alonso AM, Cottier JP, Herbreteau D. Contrast-enhanced sonography during uterine artery embolization for the treatment of leiomyomas. Ultrasound Obstet Gynecol. 2004 Jan;23(1):77-9. doi: 10.1002/uog.944. PMID 14971005